CLINICAL TRIAL: NCT00556192
Title: Can Targeted Elimination of B-cell Depletion Therapy and/or Combination Therapy Restore Peripheral B Cell Abnormalities in Systemic Lupus Erythematosus(SLE)?
Brief Title: Can Targeted Elimination of B-cell Depletion Therapy and/or Combination Therapy on Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLE-2005-006
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Rituximab; Methylprednisolone; Cyclophosphamide
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Rituximab
  Interventions: Drug: rituximab
- 2 (Active Comparator): Rituximab + Cyclophosphamide
  Interventions: Drug: rituximab
- 3 (Active Comparator): Cyclophosphamide
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 1. Rituximab of 1000 mg given 2 weeks apart. On day the of rituximab, and 'pulse' methylprednisolone 250mg IV be given followed by prednisolone 30mg/day from Day 2 to Day 5.
  2. A treatment dose rituximab of 1000mg given 2 weeks apart and 'pulse' methylprednisolone 250mg IV be given followed by prednisolone 30mg/day from Day 2 to Day 5, and 'pulse' cyclophosphamide 500mg/m2 at baseline and day 14.
  3. Sequential therapy with oral cyclophosphamide (50 to 100 mg/day) for 6 months followed by azathioprine (up to 2.5mg/kg/day) for maintenance up to 12 months. Oral prednisolone will be given at 0.5 mg/kg/day (up to 30 mg daily) for 4 weeks, tapered by 5 mg every 2 weeks thereafter until 5mg /day for the rest of the study period.
  Other Names: Mabthera

SUMMARY:
This prospective randomized control trial is undertaken to evaluate the safety and efficacy of anti-CD20 monoclonal antibody, rituximab, used as 1. monotherapy, 2. in combination with cyclophosphamide, in the treatment of proliferative lupus nephritis, as compared with standard immunosuppressive therapy with cyclophosphamide and azathioprine.

DETAILED DESCRIPTION:
Twenty patients will be randomized into 3 treatment arms to receive:

* Rituximab of 1000 mg given 2 weeks apart. On day the of rituximab, and 'pulse' methylprednisolone 250mg IV be given followed by prednisolone 30mg/day from Day 2 to Day 5.
* A treatment dose rituximab of 1000mg given 2 weeks apart and 'pulse' methylprednisolone 250mg IV be given followed by prednisolone 30mg/day from Day 2 to Day 5, and 'pulse' cyclophosphamide 500mg/m2 at baseline and day 14.
* Sequential therapy with oral cyclophosphamide (50 to 100 mg/day) for 6 months followed by azathioprine (up to 2.5mg/kg/day) for maintenance up to 12 months. Oral prednisolone will be given at 0.5 mg/kg/day (up to 30 mg daily) for 4 weeks, tapered by 5 mg every 2 weeks thereafter until 5mg /day for the rest of the study period. All patients would be started on angiotensin converting enzyme inhibitors before commencement of the trial and to continue at the same dosage throughout the study period. Patients who are on antimalarial agents and statins at baseline will be allowed to continue.

Clinical examination and laboratory investigations will be performed at 0, 4, 8, 12, 24, 36 and 48 weeks from the time of treatment. At each visit, patients will be evaluated for clinical manifestation of SLE and side effects of therapy. Laboratory parameters measured included the complete blood cell count with differential and platelet counts, chemistries survey, urinalysis, and 24- hour urinary for protein excretion and creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Active proliferative lupus nephrites
* Biopsy confirmed active proliferative lupus nephritis within 3 months prior to enrollment
* Proteinuria >= 2g/day
* Active urinary sediments
* Activity index of >= 6
* Elevated anti-double-stranded(anti-dsDNA) level at baseline
* Agreement to practice birth control
* SLE according to the American College of Rheumatology Criteria
* Informed consent was obtained

Exclusion Criteria:

* Pre-existing renal failure
* History of cancer
* Human immunodeficiency virus infection
* Active hepatitis B or C infection
* Active tuberculosis
* Diabetes mellitus
* A ny other chronic disease
* Unwillingness to comply with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
-Estimated glomerular filtration rate(FRR) of >90 mil/minute.1.73m2 -Urinary protein:urinary creatinine ratio of <0.2 -Inactive urinary sediment | wk48

SECONDARY OUTCOMES:
-The estimated GFR,urinary protein values and urinary sediment -Changes in disease activity score(SLEDAI) -Other clinical features -Duration of B-cell depletion | baseline,wk0,wk4,wk8,wk12,wk24,wk36,wk48

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Kwok Ming LI, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, China